CLINICAL TRIAL: NCT07207889
Title: Retrospective Analysis of the Efficacy of Morphine Gel (MG) for the Treatment of Pain Associated With RadioDermatitis (RD) More Than Grade II
Brief Title: Retrospective Analysis of the Efficacy of Morphine Gel to Treat Pain Associated With Perineal RadioDermatitis
Acronym: ANTAGEL
Status: Completed | Type: Observational
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Other Study IDs: DATA240316 ANTAGEL
Record Dates: First submitted 2025-08-29; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-04

CONDITIONS: Dermatitis, Radiation Induced
Keywords: morphine gel; cutaneous toxicity
MeSH Terms: conditions — Radiodermatitis | interventions — IntraSite Gel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients using morphine gel: patients who received morphine gel to treat pain due to perineal radiodermatitis
  Interventions: Drug: morphine chlorhydrate in intrasite gel

INTERVENTIONS:
Drug: morphine chlorhydrate in intrasite gel — The use of Morphine gel to treat painfull perineal radiodermatitis is new. None clinical study was conducted to explore the efficacy of the morphine gel as local analgesic for these cutaneous toxicity due to radiotherapy

SUMMARY:
Retrospective study evaluating the efficacy of a pharmacy-prepared Morphine gel used in clinics for the treatment of pain associated with perineal radiodermatitis. The main aim of this study is to evaluate the efficacy of Morphine Gel (MG) in pain management.

DETAILED DESCRIPTION:
Radiotherapy (RT) can induce acute side effects or toxicities, known as radiodermatitis (RD). Technological and technical advances have made it possible to reduce these toxicities (1), although certain organs such as the skin and mucous membranes remain vulnerable, particularly when the tumor is located nearby.

Skin exposed to ionizing radiation (IR) during the treatment of tumors close to the cutaneous surface is no longer able to renew itself due to an alteration in the basal cell mitotic process, leading to suppression of skin cell renewal. IR also induces senescence of epidermal keratinocytes, responsible for exacerbated inflammatory activity and structural dysfunction of the epidermal barrier, through disruption of the keratinization and cornification process. (2).

RD usually heals ad integrum. They are classified into 5 grades according to the Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 (3), presenting different clinical aspects ranging from grade I to V.

Grade II and III RDs are frequently observed in patients undergoing perineal RT, especially as medical treatment is associated.

In addition to the tumor's proximity to the skin, several anatomical factors specific to the perineal region contribute to the occurrence of these RDs: a wetter area, with skin folds, subject to friction and the presence of the urinary and anal orifices, potential sources of irritation by the elimination of urine and feces.

These RD are painful and have a significant impact on patients' quality of life (4,5,6). Pain intensity is often underestimated prior to treatment (7). The discomfort and pain experienced during RT intensify over the course of the sessions (8). Although RD is a frequent acute toxicity in patients treated for perineal tumors, there are few studies describing the impact of RD-related pain. The treatment of pain in RT must be rigorously assessed, and appropriate systemic or local therapy proposed (9). The challenge in treating pain in perineal radiodermatitis (PDR) is to ensure the full administration of the initial RT treatment regimen, which in the event of long interruption or premature discontinuation would expose the patient to a greater risk of recurrence (10-12).

Despite the studies carried out, there is no consensus on local care for the prevention or treatment of DR. However, the topicals used should not compromise the efficacy of RT, and should optimize healing, with gels being the preferred form.

This is why a dedicated care circuit has been set up at the Institut Curie to optimize preventive skin care and monitoring of tolerance to ROP. This system enables the early detection of painful ROP refractory to the prescribed systemic treatment.

In case of painful RD: patients are offered a hydrogel preparation mixed with morphine for local relief. Patients apply this preparation themselves during the day.

The main objective of this study is to evaluate the efficacy of morphine gel (GM) in the treatment of pain in PRD. The primary endpoint is the patient's self-reported reduction in pain. Secondary objectives include evaluation of systemic analgesic prescription and analysis of treatment interruptions attributable to DR.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years and older;
* Use of a local analgesic treatment based on Morphine gel for pain associated with perineal radiodermatitis.
* Patients not relieved by prescribed systemic treatments (per-os or intravenous)
* Patients treated with radiotherapy for a perineal tumor, whether or not associated with medical treatment such as chemotherapy.
* Minimum grade of radiodermatitis: Grade II

Exclusion Criteria:

* Patients who have not used the prescribed morphine gel
* Minor patients
* Patients using morphine gel for wounds other than radiodermatitis
* Patients who object to the re-use of their data

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 17 patients who received Morphine gel for the treatment of pain associated with perineal radiodermatitis over a 20-month period between July 2022 and March 2024.
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Efficacy of morphine gel (GM) in the treatment of pain in perineal radiodermatitis | between baseline and day2 to day21
  Reduced pain as assessed by the patient. Verbal scale to qualify the evolution of the pain (decreased - stable - increased)

SECONDARY OUTCOMES:
Assessment of systemic analgesic prescribed | between baseline and day2 to day 21
  Difference of type of non-opoïd and opioïd treatment prescribed from baseline to D2 to D21.
Interruption of radiotherapy treatment in connection with radiodermatitis | during 5 weeks from first day of radiotherapy (throught radiotherapy completion)
  Number of radiotherapy treatment breaks or discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Elodie LABEDADE, Principal Investigator — Institut Curie
Locations (1):
- Institut Curie, Paris, France